CLINICAL TRIAL: NCT03953677
Title: A Randomized Controlled Pilot Study Evaluating the Effect of Dexmedetomidine on Phenylephrine Response During Refractory Septic Shock
Brief Title: Evaluation of the Effect of Dexmedetomidine on Phenylephrine Response During Refractory Septic Shock
Acronym: Adress-Pilot
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Excess mortality in one arm of the study that led to discontinuation of enrollment
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DARGENT APJ 2018
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Septic Shock; Vasopressor Resistance
MeSH Terms: conditions — Shock, Septic | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine 100 Mcg/mL Intravenous Solution
- Placebo (Placebo Comparator)
  Interventions: Drug: 5% glucose Infusion solution

INTERVENTIONS:
Drug: Dexmedetomidine 100 Mcg/mL Intravenous Solution — Continuous infusion of dexmedetomidine at 0.7 µg/kg/h for 2 hours and then 1 µg/kg/h at fixed dose
  Arms: Dexmedetomidine
Drug: 5% glucose Infusion solution — Continuous infusion of placebo (5% glucose) at 0.7 µg/kg/h for 2 hours and then 1 µg/kg/h at fixed dose
  Arms: Placebo

SUMMARY:
Septic shock is common in patients admitted to intensive care and hospital mortality occurs in close to 50% of these patients. In half of the cases, death occurs within the first 72 hours in a context of multiple organ failure that does not respond to conventional therapies, particularly circulatory therapies, despite increasing doses of catecholamines. Vasopressor resistance in septic patients defines refractory septic shock. In one study (Conrad et al. 2015), the increase in blood pressure observed with an infusion of increasing doses of phenylephrine (dose-response curve) made it possible to quickly and clearly identify patients resistant to vasopressors at a high risk of death by refractory shock (ROC AUC 0.92). This resistance is due in particular to a downregulation of α1 adrenergic receptors, linked to sympathetic hyper activation associated with septic shock. To date, there is no validated therapy in this situation. However, experimental data have shown that the administration of α2 agonists, usually used for their sedative (dexmedetomidine) or anti-hypertensive (clonidine) effect, normalizes sympathetic activity towards basal values. In animals, α2 agonists restore the sensitivity of alpha1 adrenergic receptors, resulting in improved vasopressor sensitivity and survival. In humans, a beneficial effect on mortality was suggested in the first trial testing dexmedetomidine in septic patients in 2017. This effect was observed especially in the most severe patients, suggesting a restoration of sensitivity to vasopressors.

The hypothesis is that the administration of dexmedetomidine in patients in refractory septic shock may improve response to phenylephrine and decrease resistance to vasopressors. This pilot study could lay the foundation for a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Septic shock, defined by the "Sepsis-3" criteria

  * proven or suspected infection, with modification of the SOFA score ≥ 2 points,
  * with persistent hypotension requiring vasopressors to maintain MAP ≥ 65 mmHg
  * and a serum lactate level > 2 mmol/L despite adequate vascular filling
* Adequate vascular filling: ≥ 30ml/kg, OR absence of preload-dependency criteria at time of assessment (respiratory variability of the inferior vena cava, passive leg lift, pulsed pressure variation)
* Catecholamine resistance, defined by the need for a dose of norepinephrine ≥ 0,5 µg/kg/min for more than 2 consecutive hours within 24 hours of admission to intensive care unit
* persistence of circulatory failure with at least one of the following criteria present in the 2 hours prior to randomisation: hyperlactatemia > 2mmol/l, and/or mottling (≥ 1 score), and/or oliguria (diuresis < 0,5 ml/kg/h over the last 2 hours)
* Invasive Mechanical ventilation
* Under sedation by midazolam or propofol
* Informed consent obtained from a relative for patient included in an emergency
* Patient affiliated to the national health insurance system

Exclusion Criteria:

* Cardiac arrest before inclusion and occurring before septic shock criteria are met
* Cardiac index < 2.2 l/min/m² after volume correction, or left ventricular ejection fraction < 40% on echocardiography
* Bradycardia < 55 bpm (apart from treatment with β-blocker) or 2nd or 3rd degree BAV not equipped
* Proven or suspected decompensation of coronary heart disease
* Acute cerebrovascular condition within 2 weeks prior to inclusion
* Severe hepatic insufficiency with TP and factor V <50% in the absence of DIC (disseminated intravascular coagulation)
* Patient on adrenaline or vasopressors at the time of inclusion (epinephrine or vasopressin stopped prior to inclusion is not a criterion for non-inclusion)
* Patient on non-selective MAOI iproniazid within 15 days of inclusion
* Patient for whom a decision has been made to limit the use of therapies
* Hypersensitivity to dexmedetomidine or phenylephrine
* Patient on dexmedetomidine before inclusion
* Person subject to a legal protection measure (curatorship, guardianship)
* Person subject to limited judicial protection
* Pregnant, parturient or breastfeeding woman
* Patient with suspected or confirmed mesenteric ischemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-10-27 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Relative change in mean blood pressure, expressed as a percentage | 6 hours after the end of the initial test
  Relative variation in mean blood pressure between the basal value at the beginning of the test and the value reached at the dose of 6 µg/kg/min (%PAM0 = PAMd/PAM0 x100)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Result] Dargent A, Bourredjem A, Jacquier M, Bohe J, Argaud L, Levy B, Fournel I, Cransac A, Badie J, Quintin L, Quenot JP. Dexmedetomidine to Reduce Vasopressor Resistance in Refractory Septic Shock: alpha2 Agonist Dexmedetomidine for REfractory Septic Shock (ADRESS): A Double-Blind Randomized Controlled Pilot Trial. Crit Care Med. 2025 Apr 1;53(4):e884-e896. doi: 10.1097/CCM.0000000000006608. Epub 2025 Feb 28. PMID 40019329
- [Derived] Dargent A, Bourredjem A, Argaud L, Levy B, Fournel I, Cransac A, Badie J, Quintin L, Quenot JP. Dexmedetomidine to reduce vasopressor resistance in refractory septic shock: Protocol for a double-blind randomized controlled pilot trial (ADRESS Pilot study). Front Med (Lausanne). 2022 Aug 9;9:968274. doi: 10.3389/fmed.2022.968274. eCollection 2022. PMID 36017005